CLINICAL TRIAL: NCT00296881
Title: Clinical Outcomes Following Non-Surgical Treatment of Chronic Periodontitis, Using Scaling and Root Planing (SRP) in Conjunction With PerioWave, Compared to SRP Alone
Brief Title: SRP in Combination With PERIOWAVE in Comparison to SRP Alone in Chronic Periodontitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ondine Research Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORL-0605-3
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Periodontitis
Keywords: Periodontitis; Photodynamic Disinfection; PERIOWAVE; Scaling and Root Planing; SRP
MeSH Terms: conditions — Periodontitis

INTERVENTIONS:
Device: PERIOWAVE

SUMMARY:
This study is to determine whether scaling and root planning (SRP) followed by photodynamic disinfection results in improved outcomes that persist over time in adults with chronic periodontitis when compared with subjects with SRP alone.

DETAILED DESCRIPTION:
Extensive research has shown that lethal photosensitization with low levels of laser light is an effective method of killing numerous types of organisms. This therapy avoids the use of antibiotics along with their potential side effects. The initial application of this therapy to the oral cavity is particularly appropriate since the therapy can be applied topically either in a specific or general fashion, killing is immediate and resistance is unlikely as it is free radical-mediated. In addition, the disease states being treated (gingivitis & periodontitis) are highly prevalent and associated with significant morbidity. The equipment and costs of this therapy are simple, easily applied and relatively inexpensive compared with current therapies. Based on the scientific data to date this therapy has the potential of significantly improving the oral health of those affected.

This is a pivotal, prospective, randomized, examiner blinded, multicenter study to evaluate the effect of a single treatment of photodynamic disinfection in adults with chronic periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is capable of giving informed consent
2. Subject is willing to sign a consent form
3. Adult male or female ≥ the age of 18
4. Having been diagnosed with chronic periodontitis
5. >18 fully erupted teeth
6. Has had no periodontal instrumentation in the four months prior to the initiation of study treatment
7. Subject has at least 4 sites with pocket depth of 6-9 mm in at least two quadrants of the mouth.
8. Subject is willing and able to return for treatment and evaluation procedures scheduled throughout the course of this clinical study

Exclusion Criteria:

1. Is pregnant or nursing or who plans to become pregnant in the next 4 months
2. Having significant liver disease by subject report
3. Having an active malignancy of any type by subject report
4. Having chronic disease or diminished mental capacity that would mitigate the ability to comply with the protocol
5. Having any significant chronic disease (either acute or chronic) with concomitant oral manifestations that in the opinion of the investigator would interfere with evaluation of safety or efficacy of PerioWave®
6. Having an active periapical abscess or periodontal abscess
7. Treatment with antibiotics with in the 1-month period prior to beginning the study or any systemic condition which requires antibiotic coverage for routine periodontal procedures (e.g. heart conditions, joint replacements, etc) by report of the subject
8. History of acute necrotizing ulcerative gingivitis
9. Known allergy to Methylene Blue
10. Has glucose-6-phosphate dehydrogenase (G6PD) deficiency by subject report
11. Currently uses anti-coagulant therapy at therapeutic doses
12. Currently uses photosensitizing medications
13. Participated in investigational treatment in the last 30 days or expectation for using a separate investigational treatment during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in Periodontal Pocket Depth | 6, 12, 24, 36, 48 weeks

SECONDARY OUTCOMES:
Reduction in Bleeding on Probing | 6, 12, 24, 36, 48 weeks
Increase in Clinical Attachment Level | 6, 12, 24, 36, 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Donos, DDS, MS, PhD, Principal Investigator — University College London, Eastman Dental Institute
Locations (1):
- UCL Eastman Dental Institute, London, United Kingdom

REFERENCES:
- [Background] Albandar JM, Brunelle JA, Kingman A. Destructive periodontal disease in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):13-29. doi: 10.1902/jop.1999.70.1.13. PMID 10052767
- [Background] Brown LJ, Johns BA, Wall TP. The economics of periodontal diseases. Periodontol 2000. 2002;29:223-34. doi: 10.1034/j.1600-0757.2002.290111.x. No abstract available. PMID 12102710
- [Background] Albandar JM, Kingman A. Gingival recession, gingival bleeding, and dental calculus in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):30-43. doi: 10.1902/jop.1999.70.1.30. PMID 10052768
- [Background] Oral health in America: a report of the Surgeon General. J Calif Dent Assoc. 2000 Sep;28(9):685-95. PMID 11324049
- [Background] Socransky SS, Haffajee AD. Evidence of bacterial etiology: a historical perspective. Periodontol 2000. 1994 Jun;5:7-25. doi: 10.1111/j.1600-0757.1994.tb00016.x. No abstract available. PMID 9673160
- [Background] Haffajee AD, Socransky SS. Microbial etiological agents of destructive periodontal diseases. Periodontol 2000. 1994 Jun;5:78-111. doi: 10.1111/j.1600-0757.1994.tb00020.x. No abstract available. PMID 9673164
- [Background] Consensus report. Periodontal diseases: epidemiology and diagnosis. Ann Periodontol. 1996 Nov;1(1):216-22. doi: 10.1902/annals.1996.1.1.216. No abstract available. PMID 9118258
- [Background] Zambon JJ. Periodontal diseases: microbial factors. Ann Periodontol. 1996 Nov;1(1):879-925. doi: 10.1902/annals.1996.1.1.879. No abstract available. PMID 9118283
- [Background] Hujoel PP, Powell LV, Kiyak HA. The effects of simple interventions on tooth mortality: findings in one trial and implications for future studies. J Dent Res. 1997 Apr;76(4):867-74. doi: 10.1177/00220345970760040801. PMID 9126183
- [Background] Quirynen M, Op Heij DG, Adriansens A, Opdebeeck HM, van Steenberghe D. Periodontal health of orthodontically extruded impacted teeth. A split-mouth, long-term clinical evaluation. J Periodontol. 2000 Nov;71(11):1708-14. doi: 10.1902/jop.2000.71.11.1708. PMID 11128918
- [Background] De Soete M, Mongardini C, Peuwels M, Haffajee A, Socransky S, van Steenberghe D, Quirynen M. One-stage full-mouth disinfection. Long-term microbiological results analyzed by checkerboard DNA-DNA hybridization. J Periodontol. 2001 Mar;72(3):374-82. doi: 10.1902/jop.2001.72.3.374. PMID 11327066
- [Background] Goodson JM. Antimicrobial strategies for treatment of periodontal diseases. Periodontol 2000. 1994 Jun;5:142-68. doi: 10.1111/j.1600-0757.1994.tb00022.x. No abstract available. PMID 9673166
- [Background] Johnson V, Johnson BD, Sims TJ, Whitney CW, Moncla BJ, Engel LD, Page RC. Effects of treatment on antibody titer to Porphyromonas gingivalis in gingival crevicular fluid of patients with rapidly progressive periodontitis. J Periodontol. 1993 Jun;64(6):559-65. doi: 10.1902/jop.1993.64.6.559. PMID 8393109
- [Background] Hung HC, Douglass CW. Meta-analysis of the effect of scaling and root planing, surgical treatment and antibiotic therapies on periodontal probing depth and attachment loss. J Clin Periodontol. 2002 Nov;29(11):975-86. doi: 10.1034/j.1600-051x.2002.291102.x. PMID 12472990
- [Background] Lindhe J, Nyman S. Long-term maintenance of patients treated for advanced periodontal disease. J Clin Periodontol. 1984 Sep;11(8):504-14. doi: 10.1111/j.1600-051x.1984.tb00902.x. PMID 6384275
- [Background] Antczak-Bouckoms A, Joshipura K, Burdick E, Tulloch JF. Meta-analysis of surgical versus non-surgical methods of treatment for periodontal disease. J Clin Periodontol. 1993 Apr;20(4):259-68. doi: 10.1111/j.1600-051x.1993.tb00355.x. PMID 8473536
- [Background] Kalkwarf KL, Kaldahl WB, Patil KD. Patient preference regarding 4 types of periodontal therapy following 3 years of maintenance follow-up. J Clin Periodontol. 1992 Nov;19(10):788-93. doi: 10.1111/j.1600-051x.1992.tb02172.x. PMID 1452806
- [Background] McFall WT Jr. Tooth loss in 100 treated patients with periodontal disease. A long-term study. J Periodontol. 1982 Sep;53(9):539-49. doi: 10.1902/jop.1982.53.9.539. PMID 6957591
- [Background] Renvert S, Wikstrom M, Dahlen G, Slots J, Egelberg J. Effect of root debridement on the elimination of Actinobacillus actinomycetemcomitans and Bacteroides gingivalis from periodontal pockets. J Clin Periodontol. 1990 Jul;17(6):345-50. doi: 10.1111/j.1600-051x.1990.tb00029.x. PMID 2204636
- [Background] Sbordone L, Ramaglia L, Gulletta E, Iacono V. Recolonization of the subgingival microflora after scaling and root planing in human periodontitis. J Periodontol. 1990 Sep;61(9):579-84. doi: 10.1902/jop.1990.61.9.579. PMID 2213468
- [Background] Haffajee AD, Cugini MA, Dibart S, Smith C, Kent RL Jr, Socransky SS. Clinical and microbiological features of subjects with adult periodontitis who responded poorly to scaling and root planing. J Clin Periodontol. 1997 Oct;24(10):767-76. doi: 10.1111/j.1600-051x.1997.tb00195.x. PMID 9350562
- [Background] Niederman R, Abdelshehid G, Goodson JM. Periodontal therapy using local delivery of antimicrobial agents. Dent Clin North Am. 2002 Oct;46(4):665-77, viii. doi: 10.1016/s0011-8532(02)00030-7. PMID 12436823
- [Background] Herrera D, Sanz M, Jepsen S, Needleman I, Roldan S. A systematic review on the effect of systemic antimicrobials as an adjunct to scaling and root planing in periodontitis patients. J Clin Periodontol. 2002;29 Suppl 3:136-59; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.8.x. PMID 12787214
- [Background] Chung WO, Gabany J, Persson GR, Roberts MC. Distribution of erm(F) and tet(Q) genes in 4 oral bacterial species and genotypic variation between resistant and susceptible isolates. J Clin Periodontol. 2002 Feb;29(2):152-8. doi: 10.1034/j.1600-051x.2002.290210.x. PMID 11895543
- [Background] Wilson M, Dobson J, Harvey W. Sensitization of oral bacteria to killing by low-power laser radiation. Curr Microbiol. 1992 Aug;25(2):77-81. doi: 10.1007/BF01570963. PMID 1369193
- [Background] Malik Z, Hanania J, Nitzan Y. Bactericidal effects of photoactivated porphyrins--an alternative approach to antimicrobial drugs. J Photochem Photobiol B. 1990 May;5(3-4):281-93. doi: 10.1016/1011-1344(90)85044-w. PMID 2115912
- [Background] Martinetto P, Gariglio M, Lombard GF, Fiscella B, Boggio F. Bactericidal effects induced by laser irradiation and haematoporphyrin against gram-positive and gram-negative microorganisms. Drugs Exp Clin Res. 1986;12(4):335-42. PMID 3522156
- [Background] Dobson J, Wilson M. Sensitization of oral bacteria in biofilms to killing by light from a low-power laser. Arch Oral Biol. 1992 Nov;37(11):883-7. doi: 10.1016/0003-9969(92)90058-g. PMID 1334649
- [Background] Wilson M, Dobson J, Sarkar S. Sensitization of periodontopathogenic bacteria to killing by light from a low-power laser. Oral Microbiol Immunol. 1993 Jun;8(3):182-7. doi: 10.1111/j.1399-302x.1993.tb00663.x. PMID 8233573
- [Background] Frentzen M, Koort HJ. Lasers in dentistry: new possibilities with advancing laser technology? Int Dent J. 1990 Dec;40(6):323-32. PMID 2276829
- [Background] Sarkar S, Wilson M. Lethal photosensitization of bacteria in subgingival plaque from patients with chronic periodontitis. J Periodontal Res. 1993 May;28(3):204-10. doi: 10.1111/j.1600-0765.1993.tb01070.x. PMID 8388448
- [Background] Bhatti M, MacRobert A, Meghji S, Henderson B, Wilson M. A study of the uptake of toluidine blue O by Porphyromonas gingivalis and the mechanism of lethal photosensitization. Photochem Photobiol. 1998 Sep;68(3):370-6. PMID 9747591
- [Background] Dougherty TJ, Grindey GB, Fiel R, Weishaupt KR, Boyle DG. Photoradiation therapy. II. Cure of animal tumors with hematoporphyrin and light. J Natl Cancer Inst. 1975 Jul;55(1):115-21. doi: 10.1093/jnci/55.1.115. PMID 1159805
- [Background] Paardekooper M, Van den Broek PJ, De Bruijne AW, Elferink JG, Dubbelman TM, Van Steveninck J. Photodynamic treatment of yeast cells with the dye toluidine blue: all-or-none loss of plasma membrane barrier properties. Biochim Biophys Acta. 1992 Jul 8;1108(1):86-90. doi: 10.1016/0005-2736(92)90117-5. PMID 1322699
- [Background] Paardekooper M, De Bruijne AW, Van Steveninck J, Van den Broek PJ. Inhibition of transport systems in yeast by photodynamic treatment with toluidine blue. Biochim Biophys Acta. 1993 Sep 19;1151(2):143-8. doi: 10.1016/0005-2736(93)90097-j. PMID 8373789
- [Background] Paardekooper M, De Bruijne AW, Van Steveninck J, Van den Broek PJ. Intracellular damage in yeast cells caused by photodynamic treatment with toluidine blue. Photochem Photobiol. 1995 Jan;61(1):84-9. doi: 10.1111/j.1751-1097.1995.tb09247.x. PMID 7899497
- [Background] Wilson M, Mia N. Sensitisation of Candida albicans to killing by low-power laser light. J Oral Pathol Med. 1993 Sep;22(8):354-7. doi: 10.1111/j.1600-0714.1993.tb01088.x. PMID 7506775
- [Background] Smetana Z, Ben-Hur E, Mendelson E, Salzberg S, Wagner P, Malik Z. Herpes simplex virus proteins are damaged following photodynamic inactivation with phthalocyanines. J Photochem Photobiol B. 1998 Jun 15;44(1):77-83. doi: 10.1016/S1011-1344(98)00124-9. PMID 9745730
- [Background] Position paper: epidemiology of periodontal diseases. American Academy of Periodontology. J Periodontol. 1996 Sep;67(9):935-45. PMID 8884652
- [Background] Birch JF, Mandley DJ, Williams SL, Worrall DR, Trotter PJ, Wilkinson F, Bell PR. Methylene blue based protein solder for vascular anastomoses: an in vitro burst pressure study. Lasers Surg Med. 2000;26(3):323-9. doi: 10.1002/(sici)1096-9101(2000)26:33.0.co;2-r. PMID 10738296
- [Background] Luksiene Z. Photodynamic therapy: mechanism of action and ways to improve the efficiency of treatment. Medicina (Kaunas). 2003;39(12):1137-50. PMID 14704501
- [Background] O'Neill J, Wilson M, Wainwright M. Comparative antistreptococcal activity of photobactericidal agents. J Chemother. 2003 Aug;15(4):329-34. doi: 10.1179/joc.2003.15.4.329. PMID 12962360
- [Background] Wainwright M. Photodynamic antimicrobial chemotherapy (PACT). J Antimicrob Chemother. 1998 Jul;42(1):13-28. doi: 10.1093/jac/42.1.13. PMID 9700525
- [Background] Bertoloni G, Zambotto F, Conventi L, Reddi E, Jori G. Role of specific cellular targets in the hematoporphyrin-sensitized photoinactivation of microbial cells. Photochem Photobiol. 1987 Nov;46(5):695-8. doi: 10.1111/j.1751-1097.1987.tb04834.x. No abstract available. PMID 3327061
- [Background] Bhatti M, Nair SP, Macrobert AJ, Henderson B, Shepherd P, Cridland J, Wilson M. Identification of photolabile outer membrane proteins of Porphyromonas gingivalis. Curr Microbiol. 2001 Aug;43(2):96-9. doi: 10.1007/s002840010268. PMID 11391471